CLINICAL TRIAL: NCT04884607
Title: Electrocardiogram Measurement and Subthreshold Low-level Autonomic Nerve Stimulation Using External Auditory Canal Electrodes
Brief Title: Autonomic Nerve Stimulation Using External Auditory Canal Electrodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seil Oh, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-2104-191-1214
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Arrhythmia; Cardiovascular Diseases
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Study group will receive subthreshold low-level autonomic nerve stimulation using external auditory canal electrodes.
  Interventions: Other: subthreshold low-level autonomic nerve stimulation using external auditory canal electrodes

INTERVENTIONS:
Other: subthreshold low-level autonomic nerve stimulation using external auditory canal electrodes — * Evaluation of electrocardiogram measurement from external auditory canal electrodes: Participants are required to attach specially designed external auditory canal electrodes to their both ears to record electrocardiogram. Both electrocardiogram from the precordium and the ear would be simultaneously recorded and compared.
  * Evaluation of low-level autonomic nerve stimulation using external auditory canal: Using the electrodes described above, Arnold's nerve will be stimulated with low-level electric impulses using TENS device. During and after the stimulation, heart rate variability will be measured to investigate the impact of nerve stimulation on autonomic function modulation on the heart.

SUMMARY:
* Purpose of the study This study aimed to investigate electrocardiogram measurement and subthreshold low-level autonomic nerve stimulation using external auditory canal electrodes among healthy adult participants
* Study design Prospective, single-center, interventional, single-arm design
* Study participants A total of 12 healthy adult participants without cardiovascular diseases will be recruited.
* Study methods

  1. Participant enrollment Study participants will be recruited by advertisement posters announced at the lobby of the hospital
  2. Evaluation of electrocardiogram measurement from external auditory canal electrodes Participants are required to attach specially designed external auditory canal electrodes to their both ears to record electrocardiogram. Both electrocardiogram from the precordium and the ear would be simultaneously recorded and compared.
  3. Evaluation of low-level autonomic nerve stimulation using external auditory canal Using the electrodes described above, Arnold's nerve will be stimulated with low-level electric impulses using TENS device. During and after the stimulation, heart rate variability will be measured to investigate the impact of nerve stimulation on autonomic function modulation on the heart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults without cardiovascular diseases
* Aged 20 years or more with Informed consent

Exclusion Criteria:

* Patients with autonomic disorder, cardiovascular drug prescriptions, cardiovascular diseases, diabetes, or with cardiac implantable electronic devices
* Patients with abnormalities at both external auditory canals and ears

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Through study completion, an average of within 1 day
  Selected parameters of heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Seil Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available upon appropriateness of the request.